CLINICAL TRIAL: NCT03953508
Title: Menthol and Non-Menthol Cigarette Smoking in Young Adults
Brief Title: Perceptions of Cigarette Smoking in Young Adults
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRISM
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol (Other): Participants who prefer smoking menthol cigarettes
  Interventions: Other: Cigarette flavor type
- Non-menthol (Other): Participants who prefer smoking non-menthol cigarettes
  Interventions: Other: Cigarette flavor type

INTERVENTIONS:
Other: Cigarette flavor type — Participants will smoke several puffs (each) of a menthol Camel Crush and several puffs of a non-menthol Camel Crush cigarette.
  Other Names: Experimental cigarette smoking

SUMMARY:
This study focuses on menthol (n = 125) and non-menthol (n = 125) smoking young adults (YAs; defined here as ages 18 to 26).

DETAILED DESCRIPTION:
The study will occur in three phases.

In session 1 of Phase 1, participants will engage in ad libitum smoking session of one's preferred cigarette brand (menthol or non-menthol). In session 2, participants will take several puffs each of a commercially available menthol and non-menthol cigarette (i.e., Camel Crush) and complete a complete a series of pre-post smoking questionnaires, and in Session 3 participants will complete a computerized task to measure perceptions of cigarette smoking. For the computerized task, participants will be able to "win" points toward earning puffs of a cigarette and will be able to smoke puffs earned. Participants will be asked to abstain from smoking for at least 12 hours before each in-person visit.

Phase 2 participants will engage in 14 days of surveys they will complete on their cell to measure different aspects of smoking behavior. These surveys will happen twice a day at random times.

For phase 3, participants will complete an assessment of smoking behavior and related factors 6-months after the baseline assessment either in-person, in the laboratory, or via telephone or online (if in-person follow-up is not viable).

The order in which phases occur differed was a result of COVID-19 restrictions on data collection. For some participants, they started EMA first and then began laboratory data collection when in-person was allowed. For others, they started laboratory data collection when COVID restrictions were lifted. Thus, the participant flow may appear unbalanced.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-26
* Currently smoke cigarettes "everyday" or "somedays"
* A strong preference for menthol or non-menthol cigarettes
* able to read and understand the consent form
* willingness to abstain from nicotine or tobacco products for at least 12 hours prior to smoking sessions

Exclusion Criteria:

* Current use of nicotine replacement therapy
* Pregnant or planning to become pregnant; or breastfeeding
* self-reported diagnosis of lung disease, including asthma, cystic fibrosis, or chronic obstructive pulmonary disease; or
* self-reported history of cardiac event or distress within the past 3-months

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cohn, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohn AM, Elmasry H, Niznik T, Pickworth W, Smith MA, Margaritis WD, Wyatt R, Dunn D, Hedeker D, Murphy J, Audrain-McGovern J, Villanti AC. Racial and ethnic differences in topography and subjective effects among young adults in response to smoking their usual brand menthol or nonmenthol cigarette. Exp Clin Psychopharmacol. 2025 Apr;33(2):145-154. doi: 10.1037/pha0000765. Epub 2025 Feb 24. PMID 39992758
- [Derived] Cohn AM, Pickworth W, Audrain-McGovern J, Murphy J, Villanti AC, Hedeker D, Dunn D, Wyatt R, Niznik T, Cotten W, Smith M, Ehlke SJ. Measuring young adult appeal for menthol and non-menthol cigarettes: protocol of a clinical trial using both laboratory and intensive longitudinal methods (PRISM). BMJ Open. 2022 Apr 28;12(4):e058823. doi: 10.1136/bmjopen-2021-058823. PMID 35487522

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The order in which phases occurred differed as a result of COVID-19 restrictions on in-person data collection. Some participants started EMA first and then began laboratory data collection when in-person data collection was allowed. Other participants started laboratory data collection first (when COVID restrictions were lifted), and then did EMA after laboratory data collection. Thus, the participant flow may appear unbalanced.
Groups:
- Menthol Status: Those who prefer menthol cigarettes
- Non-menthol Status: Those who prefer non-menthol
Period: Baseline
Arm/Group | Menthol Status | Non-menthol Status
Started (The order in which phases occurred differed as a result of COVID-19 restrictions on in-person data collection. Some participants started EMA first and then began laboratory data collection when in-person data collection was allowed. Other participants started laboratory data collection first (when COVID restrictions were lifted), and then did EMA after laboratory data collection. Thus, the participant flow may appear unbalanced.) | 95 | 104
Completed | 92 | 102
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2
Period: Ecological Momentary Assessment
Arm/Group | Menthol Status | Non-menthol Status
Started (The order in which phases occurred differed was a result of COVID-19 restrictions on data collection. For some participants, they started EMA first and then began laboratory data collection when in-person was allowed. For others, they started laboratory data collection when COVID restrictions were lifted, and then did EMA. Thus, the participant flow may appear unbalanced.) | 65 | 74
Completed | 63 | 62
Not Completed | 2 | 12
Period: Laboratory Period
Arm/Group | Menthol Status | Non-menthol Status
Started (The order in which phases occurred differed was a result of COVID-19 restrictions on data collection. For some participants, they started EMA first and then began laboratory data collection when in-person was allowed. For others, they started laboratory data collection when COVID restrictions were lifted, and then did EMA. Thus, the participant flow may appear unbalanced.) | 59 | 59
Completed | 54 | 54
Not Completed | 5 | 5
Period: 6-month Follow-up
Arm/Group | Menthol Status | Non-menthol Status
Started | 92 (The number started is based on the number who completed baseline. These are the individuals who were eligible to start a follow-up.) | 102 (The number started is based on the number who completed baseline. These are the individuals who were eligible to start a follow-up.)
Completed | 30 | 32
Not Completed | 62 | 70
Not completed — Lost to Follow-up | 62 | 70

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the baseline survey and attended the first study session to smoke their usual brand cigarette. Some participants completed the baseline survey remotely, due to COVID, and then came to the laboratory to complete the first study visit. Not everyone who completed the baseline survey remotely showed up for the first study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Menthol Status | Non-menthol Status | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (2.2) | 24.2 (2.0) | 23.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 24 | 28 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 39 | 76
  Non-White | 23 | 22 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 61 | 121
Highest level of education [Count of Participants; unit: Participants]
  High school education or less | 24 | 35 | 59
  Some college education or more | 36 | 26 | 62
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 8.1 (5.4) | 11.8 (7.4) | 10 (6.7)
Past 30-day cigarette smoking frequency [Mean (Standard Deviation); unit: Number of days smoked cigarettes] | 24.0 (8.7) | 26.5 (7.9) | 25.2 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Response to Smoking Cigarettes From the Cigarette Evaluation Scale
Description: ratings of subjective satisfaction from smoking cigarettes, 1= not at all to 7 = extremely. Higher scores indicate greater positive subjective response. The minimum score is 1and the maximum score is 7.
Time Frame: immediately after smoking usual brand cigarette, at baseline
Population: Young adult menthol and non-menthol smokers, ages 18-26 who completed the baseline/first study visit
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Menthol; Non-menthol: Participants will smoke and rate puffs of their preferred brand/flavor cigarette.
Arm/Group | Menthol | Non-menthol
Number analyzed (Participants) | 60 | 61
score on a scale | 4.68 (0.16) | 4.50 (0.16)
Statistical Analysis 1: Comparison: Menthol vs Non-menthol; Test type: Other — Analysis of covariance test; p > .05, ANCOVA — Threshold for significance is p<.05

2. Primary Outcome: Average Daily Subjective Response From Smoking
Description: average daily scores of subjective reward from smoking from daily diary surveys, 1= not at all to 7 = extremely. Higher scores indicate greater positive subjective response. Averaged across 14 days.
Time Frame: Phase 2 daily diary surveys (estimated 2-4 weeks after baseline)
Population: Young adult menthol and non-menthol smokers who reported on their daily cigarette smoking during 14-days of ecological momentary assessment
Measure: Mean (Standard Deviation); unit: average daily scores
Groups:
- Most Recent Cigarette Was Non-menthol: The most recent cigarette smoked was non-menthol
- Most Recent Cigarette Was Menthol: The most recent cigarette smoked was menthol
Arm/Group | Most Recent Cigarette Was Non-menthol | Most Recent Cigarette Was Menthol
Number analyzed (Participants) | 62 | 62
average daily scores | 1.68 (0.98) | 1.79 (0.86)
Statistical Analysis 1: Comparison: Most Recent Cigarette Was Non-menthol vs Most Recent Cigarette Was Menthol; Test type: Other — T-test comparing differences, the null hypothesis is that the groups are equal; p > .05, t-test, 2 sided — Threshold for significance is p<.05

3. Primary Outcome: Highest Trial Competed for a Menthol Cigarette Puff in the Choice Task (Relative Reinforcing Value for Menthol Cigarettes)
Description: Participants completed a choice task assessing willingness to "work" to click targets on a computer screen to earn menthol or non-menthol cigarette puffs. The relative reinforcing value for menthol was defined by the Breakpoint, or the highest trial (out of 10 trials) completed for a menthol cigarette puff.
Time Frame: Lab session 3 (estimated average 1-4 weeks after baseline)
Population: young adult cigarette smokers ages 18-26 who completed the third of three laboratory sessions
Measure: Mean (Standard Deviation); unit: highest trial competed for menthol puffs
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 54 | 53
highest trial competed for menthol puffs | 9.2 (2.05) | 0.83 (2.47)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — Analysis of variance test comparing average breakpoint for menthol and non-menthol smokers; p < .05, ANOVA — Threshold for significance is p<.05

4. Primary Outcome: Past 30-day Cigarette Smoking Frequency
Description: Number of days smoked cigarettes in the past 30-days
Time Frame: 6-month follow-up survey (6-months post-baseline)
Population: Young adult smokers ages 18-26 who completed the 6-month follow-up survey
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 24 | 31
days | 20.8 (11.9) | 20.7 (11.4)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — T-test; p < .05, t-test, 2 sided — Threshold for significance is p<.05

5. Primary Outcome: Puff Topography
Description: Number of cigarette puffs after smoking one's preferred brand/flavor during lab session 1, Phase 1.
Time Frame: Laboratory session 1 (up to 4 weeks after baseline)
Population: young adult cigarette smokers ages 18-26 who completed the baseline/visit 1 and provided valid puff topography data
Measure: Mean (Standard Deviation); unit: number of cigarette puffs
Groups:
- Menthol; Non-menthol: Participants who smoked puffs of their preferred brand/flavor cigarette.
Arm/Group | Menthol | Non-menthol
Number analyzed (Participants) | 60 | 61
number of cigarette puffs | 18.7 (6.1) | 18.4 (7.3)
Statistical Analysis 1: Comparison: Menthol vs Non-menthol; Test type: Other — Analysis of variance; p > .05, ANOVA — Threshold for significance is p<.05

6. Secondary Outcome: Number of Clicks for Menthol Cigarette Puffs on the Behavioral Choice Task
Description: This outcome represents the total number of clicks (over 10 trials) for the menthol cigarette puff on the behavioral choice task. The reinforcement schedule to click/earn a menthol cigarette puff increased progressively by 25 clicks at each trial such that 25, 50, 75, 100, 125, 150, 175, 200, 225, and 250 clicks of the menthol cigarette image on a computer screen had to be achieved to earn a menthol puff at each trial (maximum possible of 1375 clicks over the task for menthol puffs). All puffs were taken once the entire task was completed (after all 10 trials were done).
Time Frame: immediately after completing the behavioral economic choice task, lab session 3 (estimated average 1-4 weeks after baseline)
Population: Young adult cigarette smokers (ages 18-26) who completed session 3
Measure: Mean (Standard Deviation); unit: number of clicks for menthol puffs
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 54 | 53
number of clicks for menthol puffs | 1244.56 (326.49) | 104.11 (334.44)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — Analysis of variance; p < .05, ANOVA — Threshold for significance is p<.05

7. Secondary Outcome: Quantity of Past 30-day Tobacco Product Use
Description: Number of tobacco products used in the past 30-days
Time Frame: 6-month follow-up (6-months post-baseline)
Population: Young adult smokers ages 18-26
Measure: Mean (Standard Deviation); unit: tobacco products
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 24 | 31
tobacco products | 1.3 (1) | 2 (0.9)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — T-test; p < .05, t-test, 2 sided — Threshold for significance is p<.05

8. Secondary Outcome: Number of Participants With Intentions to Smoke Menthol Cigarettes
Description: Number of participants who self-reported intentions to smoke menthol cigarettes assessed via a questionnaire
Time Frame: 6-month follow-up (6-months post-baseline)
Population: Young adult cigarette smokers ages 18-26
Measure: Count of Participants; unit: Participants
Groups:
- Non-menthol Smokers at the 6-month Follow-up: Those who did not reporting using any menthol cigarettes in the past 30-days at the 6-month follow-up
Arm/Group | Non-menthol Smokers at the 6-month Follow-up
Number analyzed (Participants) | 20
Participants | 16
Statistical Analysis 1: Comparison: Non-menthol Smokers at the 6-month Follow-up; Test type: Other — Fisher's exact test; p > .05, Fisher Exact — Threshold for significance is p<.05

9. Secondary Outcome: Cigarettes Per Day
Description: Daily report of numbers of cigarettes smoked per day, over 14 days
Time Frame: Phase 2 daily diary surveys (estimated 2-4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 62 | 62
cigarettes per day | 9.9 (7.6) | 9.5 (7.6)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — T-test; p > .05, t-test, 2 sided — Threshold for significance is p<.05

10. Secondary Outcome: Average Daily Craving From Smoking
Description: Average daily cigarette craving, aggregated over 14 days, from a 1-item questionnaire measure that was administered daily. Scores range from 0 = not at all to 4 = extremely, where higher scores indicate greater craving intensity.
Time Frame: Phase 2 daily diary surveys (estimated 2-4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: average daily scores
Arm/Group | Menthol Status | Non-menthol Status
Number analyzed (Participants) | 62 | 62
average daily scores | 1.55 (0.75) | 1.53 (0.75)
Statistical Analysis 1: Comparison: Menthol Status vs Non-menthol Status; Test type: Other — T-test; p > .05, t-test, 2 sided — Threshold for significance is p<.05

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the entirety of study participation; approximately 6 months.
Description: One participant vomited after smoking a cigarette in the study lab, after smoking a non-menthol Camel Crush cigarette. The participant was instructed to smoke 3 to 5 puffs In a subsequent follow-up (approximately a week later), the participant was feeling fine and wanted to schedule their next session. The participant indicated that they thought they had food poisoning. The adverse event was reported to the IRB and was not considered due to enrollment in the study or the study procedures.
Arm/Group | Menthol Status | Non-menthol Status
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 1/61
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menthol Status (N=60) | Non-menthol Status (N=61)
Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Participant vomited after smoking a study cigarette in the laboratory.

LIMITATIONS AND CAVEATS:
Data were collected during the COVID-19 pandemic, during times when there were complete or intermittent shut-downs in-person data collection. This resulted in some changes to the order of administration of the study periods/phases in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT03953508/Prot_SAP_000.pdf